CLINICAL TRIAL: NCT00967330
Title: A Study of Avastin (Bevacizumab) and Irinotecan Versus Temozolomide Radiochemistry in Patients With Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21965; 2009-010390-21
Record Dates: First submitted 2009-06-16; First posted 2009-08-27 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Irinotecan; Temozolomide

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: irinotecan
- 2 (Active Comparator)
  Interventions: Drug: temozolomide

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 10mg/kg iv every 2 weeks
  Arms: 1
Drug: irinotecan — 125mg/m2 iv every 2 weeks
  Arms: 1
Drug: temozolomide — 75mg/m2 po daily during radiotherapy, followed by 150-200mg/m2/day po on days 1-5 of each 6x4 week cycle of adjuvant therapy
  Arms: 2

SUMMARY:
This 2 arm study will compare the effect of Avastin + irinotecan versus temozolomide, in combination with conventional involved field radiotherapy, in patients with newly diagnosed glioblastoma and a non-methylated MGMT promoter. Patients will be randomized 3:1 to receive Avastin 10mg/kg iv every 2 weeks + irinotecan 125mg/m2 iv every 2 weeks, or temozolomide 75mg/m2 po daily during radiotherapy followed by 6 cycles of temozolomide 150-200mg/m2 po daily on days 1-5 of each 4 week cycle. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-70 years of age;
* glioblastoma, confirmed histologically;
* no previous chemotherapy or radiotherapy for glioblastoma;
* non-methylated MGMT promoter in the tumor.

Exclusion Criteria:

* prior systemic treatment for glioblastoma multiforme;
* prior treatment with Avastin;
* significant cardiovascular disease;
* other active malignant disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Germany (23):
  - Aachen
  - Berlin
  - Bochum
  - Bonn
  - Chemnitz
  - Cologne
  - Dresden
  - Düsseldorf
  - Erfurt
  - Erlangen
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Göttingen
  - Idar-Oberstein
  - Kiel
  - Leipzig
  - Mannheim
  - Marburg
  - München
  - Münster
  - Regensburg
  - Tübingen
  - Ulm

REFERENCES:
- [Derived] Schafer N, Proescholdt M, Steinbach JP, Weyerbrock A, Hau P, Grauer O, Goldbrunner R, Friedrich F, Rohde V, Ringel F, Schlegel U, Sabel M, Ronellenfitsch MW, Uhl M, Grau S, Hanel M, Schnell O, Krex D, Vajkoczy P, Tabatabai G, Mack F, Schaub C, Tzaridis T, Niessen M, Kebir S, Leutgeb B, Urbach H, Belka C, Stummer W, Glas M, Herrlinger U. Quality of life in the GLARIUS trial randomizing bevacizumab/irinotecan versus temozolomide in newly diagnosed, MGMT-nonmethylated glioblastoma. Neuro Oncol. 2018 Jun 18;20(7):975-985. doi: 10.1093/neuonc/nox204. PMID 29121274
- [Derived] Herrlinger U, Schafer N, Steinbach JP, Weyerbrock A, Hau P, Goldbrunner R, Friedrich F, Rohde V, Ringel F, Schlegel U, Sabel M, Ronellenfitsch MW, Uhl M, Maciaczyk J, Grau S, Schnell O, Hanel M, Krex D, Vajkoczy P, Gerlach R, Kortmann RD, Mehdorn M, Tuttenberg J, Mayer-Steinacker R, Fietkau R, Brehmer S, Mack F, Stuplich M, Kebir S, Kohnen R, Dunkl E, Leutgeb B, Proescholdt M, Pietsch T, Urbach H, Belka C, Stummer W, Glas M. Bevacizumab Plus Irinotecan Versus Temozolomide in Newly Diagnosed O6-Methylguanine-DNA Methyltransferase Nonmethylated Glioblastoma: The Randomized GLARIUS Trial. J Clin Oncol. 2016 May 10;34(14):1611-9. doi: 10.1200/JCO.2015.63.4691. Epub 2016 Mar 14. PMID 26976423

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Irinotecan: In the Concurrent Phase participants received radiotherapy in daily fractions of 1.8 to 2 Gray (Gy) given 5 fractions per week for 6 to 7 weeks and intravenous infusion (IV) of bevacizumab (BEV) 10 milligrams per kilogram (mg/kg) body weight every 14 ± 2 days starting during the first week to the last week of radiotherapy. Participants then entered the Maintenance Phase where they received BEV 10 mg/kg body weight and IV irinotecan (IRI) 125 milligrams per square meter (mg/m^2) body surface area (BSA) or 340 mg/m^2 BSA in participants not receiving enzyme-inducing antiepileptic drugs (EIAEDs) or receiving EIAEDs, respectively for every 14± 2 days until progressive disease (PD) or for a maximum treatment period of 2 years after inclusion of the last participant.
- Temozolomide: In the Concurrent Phase participants received radiotherapy in daily fractions of 1.8 to 2 Gy given 5 fractions per week for 6 to 7 week and temozolomide (TMZ) capsule 75 mg/m^2 BSA daily from the first day to the last day of radiotherapy . There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of TMZ 150 to 200 mg/m^2 BSA daily in the first 5 days of each cycle until PD or for a maximum treatment period of 2 years after inclusion of the last participant. Only participants with progressive disease during or after TMZ therapy could receive bevacizumab (BEV)/irinotecan (IRI) or BEV monotherapy as optional second-line study therapy at the discretion of the investigator, if eligible.
Period: Overall Study
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Started | 122 | 60
Completed | 0 | 0
Not Completed | 122 | 60
Not completed — Protocol Violation | 3 | 4
Not completed — Regular | 10 | 3
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Death | 102 | 51
Not completed — Severe protocol deviation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The randomized (RND) population was defined to include all participants randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Irinotecan | Temozolomide | Total
Number analyzed (Participants) | 122 | 60 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.17) | 56.4 (10.84) | 55.7 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 21 | 60
  Male | 83 | 39 | 122

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Progression-Free Survival (PFS) Without Disease Progression or Death at 6 Months
Description: Progression-free survival was defined as the time from randomization to objective tumor progression or death from any cause, whichever came first. Progression was defined as 25 percent (%) increase in size of enhancing tumor or any new tumor on gadolinium contrast agent magnetic resonance imaging (Gd-MRI) scans, or neurologically worse, and steroids stable or increased. Percentage of participants achieving PFS without disease progression or death was reported.
Time Frame: 6 months
Population: Intent-to-treat (ITT) population included participants randomized for whom it cannot be ruled out, that they took study medication at least once and where primary variable was measured at least once under study medication. Data were analyzed according to the treatment randomized (as randomized).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
percentage of participants | 79.31 [68.859 to 84.617] | 42.59 [26.680 to 53.050]
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was defined as the time from randomization to objective tumor progression or death from any cause, whichever came first. Progression was defined as 25% increase in size of enhancing tumor or any new tumor on Gd-MRI scans, or neurologically worse, and steroids stable or increased. PFS was estimated using Kaplan-Meier method.
Time Frame: From baseline to the end of the study (up to 4.5 years)
Population: ITT population. Data were analyzed according to the treatment randomized (as randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
Months | 9.74 [8.72 to 10.76] | 5.99 [2.73 to 6.15]
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Test type: Superiority or Other; p = 0.0012, Chi-squared; Hazard Ratio (HR) = 0.588, 95% CI 2-sided [0.423 to 0.817]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to death from any cause. OS was estimated using Kaplan-Meier method.
Time Frame: From baseline until death (up to 4.5 years)
Population: ITT population. Data were analyzed according to the treatment randomized (as randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
Months | 16.64 [15.43 to 18.36] | 17.30 [14.77 to 20.36]
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Test type: Superiority or Other; p = 0.8283, Chi-squared; Hazard Ratio (HR) = 0.963, 95% CI 2-sided [0.684 to 1.354]

4. Secondary Outcome: Percentage of Participants Who Discontinued
Description: Discontinuation was defined as the percentage of participants who permanently discontinued treatment in either treatment arm. Percentage of participant with individual discontinuation reason are reported. CNS: central nervous system; CTCAE: Common Terminology Criteria for Adverse Events . Other reason refers to any other reason than the specified ones.
Time Frame: From baseline until death (up to 4.5 years)
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
percentage of participants
  Persisting non-hematological toxicity CTCAE Grade3 | 0 | 1.9
  CNS hemorrhagic event (CTCAE Grade >1) | 0.9 | 0
  Gastro-intestinal perforation (CTCAE Grade 1-4) | 0.9 | 0
  Other | 9.5 | 5.6
  Participant's wish | 6 | 5.6
  Progressive disease | 74.1 | 57.4
  Proteinuria (nephrotic syndrome) (CTCAE Grade 4) | 0.9 | 0
  Regular | 1.7 | 27.8
  Repeated CTCAE Grade 4 hematological toxicity | 0 | 0.9
  Venous thrombosis/embolism | 0.9 | 0
  Wound dehiscence requiring medical intervention | 0.9 | 0
  Wound dehiscence requiring surgical intervention | 4.3 | 0

5. Secondary Outcome: Number of Participants With A Best Overall Response (BOR) of Complete Response (CR) and With A BOR of CR or Partial Response (PR)
Description: BOR was defined as the best response observed for a participant during assessment. Number of participants who had BOR as CR and number of participants who had BOR as CR or PR were reported. Complete response was defined as disappearance of all enhancing tumor on consecutive Gd-MRI scans at least 1 month apart, off steroids, and neurologically stable or improved. Partial response was defined as 50% reduction in size of enhancing tumor on consecutive Gd-MRI scans at least 1 month apart, steroids stable or reduced, and neurologically stable or improved.
Time Frame: 4 week after radiotherapy (RT) (up to Week 4), >4 Week after RT (up to Week 8) and Month 6
Population: ITT population. Data were analyzed according to the treatment randomized (as randomized). Here, number of participants analyzed = participants who were evaluable for this outcome and n = participants who were evaluable of specified time-point.
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 110 | 46
participants
  CR at 4 weeks after RT (n=110,46) | 11 | 2
  CR at >4 weeks after RT (n=95,35) | 11 | 1
  CR at Month 6 (n=91,28) | 3 | 1
  CR or PR at 4 Week after RT (n=110,46) | 42 | 6
  CR or PR at >4 Week after RT (n=95,35) | 18 | 3
  CR or PR at Month 6 (n=91,28) | 5 | 3
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Response rate based on participants with CR at 4 weeks after RT; Test type: Superiority or Other; p = 0.34745, Fisher Exact; Difference in response rate = 0.06, 95% CI 2-sided [-0.02 to 0.14]
Statistical Analysis 2: Comparison: Bevacizumab + Irinotecan vs Temozolomide; The response rate based on participants with CR at >4 weeks after RT; Test type: Superiority or Other; p = 0.17923, Fisher Exact; Difference in response rate = 0.09, 95% CI 2-sided [0.00 to 0.17]
Statistical Analysis 3: Comparison: Bevacizumab + Irinotecan vs Temozolomide; The response rate based on participants with CR at Month 6; Test type: Superiority or Other; p = 1.00000, Fisher Exact; Difference in response rate = -0.00, 95% CI 2-sided [-0.08 to 0.08]
Statistical Analysis 4: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Response rate based on participants with CR or PR at 4 weeks after RT; Test type: Superiority or Other; p = 0.00210, Fisher Exact; Difference in response rate = 0.25, 95% CI 2-sided [0.12 to 0.38]
Statistical Analysis 5: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Response rate based on participants with CR and PR at >4 weeks after RT; Test type: Superiority or Other; p = 0.18761, Fisher Exact; Difference in response rate = 0.10, 95% CI 2-sided [-0.02 to 0.23]
Statistical Analysis 6: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Response rate based on participants with CR or PR at Month 6; Test type: Superiority or Other; p = 0.38974, Fisher Exact; Difference in response rate = -0.05, 95% CI 2-sided [-0.18 to 0.07]

6. Secondary Outcome: Percentage of Participants With Response on FLAIR Imaging
Description: FLAIR lesions were determined as "stable", "progressive" or "decreased". FLAIR lesions was determined as "progressive" only if they were not be attributed to causes apart from tumor infiltration (sequelae of radiation therapy, demyelination, ischemia, infection, seizures, or other treatment effects). Percentage of participants are based on ITT population.
  Dis.=Discontinuation.
Time Frame: At screening, Baseline, Month 6 and Therapy Discontinuation (Up to 4.5 years)
Population: ITT population. Here, n = participants with at least 1 assessment during specified time-point.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
percentage of participants
  Screening: Initial Flair Lesion (n=116,54) | 72.4 | 72.2
  Screening:Stable Flair Lesion (n=116,54) | 17.2 | 16.7
  Baseline:Decreased FLAIR Lesions (n=105,46) | 16.4 | 20.4
  Baseline:Initial FLAIR Lesions (n=105,46) | 18.1 | 18.5
  Baseline:Progressive FLAIR Lesions (n=105,46) | 14.7 | 11.1
  Baseline: Stable FLAIR Lesions (n=105,46) | 41.4 | 35.2
  Month 6:Progressive FLAIR Lesions (n=91,28) | 16.4 | 22.2
  Month 6: Stable FLAIR Lesions (n=91,28) | 62.1 | 29.6
  Therapy Dis.:Decreased FLAIR Lesions (n=55,31) | 0.9 | 0.0
  Therapy Dis.:Progressiv FLAIR Lesions (n=55,31) | 29.3 | 27.8
  Therapy Dis.:Stable FLAIR Lesions (n=55,31) | 17.2 | 29.6

7. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ - C30) at Baseline, Post-Baseline (up to Month 30)
Description: The EORTC QLQ-C30 incorporates: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties); and a global health and quality-of-life scale. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores were averaged and transformed to 0-100 scale; higher score for Global Qol/functional scales=better level of functioning or a higher score for symptom scale=greater degree of symptoms. The change in global health status was determined to be the difference in values at baseline and each specific visit. The term ''baseline'' refers to the time of randomization to the maintenance phase.
Time Frame: Baseline, Post-Baseline (up to Month 30)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
units on a scale
  Physical Functioning | -8.3513 [-11.8714 to -4.8312] | -6.2511 [-11.2130 to -1.2892]
  Role Functioning | -0.7635 [-6.1695 to 4.6425] | -2.2339 [-9.9836 to 5.5159]
  Emotional Functioning | 2.2774 [-1.7409 to 6.2958] | 2.2547 [-3.4834 to 7.9928]
  Cognitive Functioning | -2.0188 [-6.2256 to 2.1880] | -3.8401 [-9.8118 to 2.1317]
  Social Functioning | -6.2324 [-11.3480 to -1.1169] | -4.6198 [-11.9009 to 2.6613]
  Global health Status /QoL (ql) | -3.1134 [-6.5412 to 0.3145] | 0.3855 [-4.4220 to 5.1930]
  Fatique | 5.5228 [1.6424 to 9.4031] | 2.1779 [-3.3223 to 7.6781]
  Nausea/Vomitting | 8.9557 [6.5139 to 11.3974] | 4.7597 [1.3958 to 8.1235]
  Pain | 10.6876 [5.8004 to 15.5747] | 1.5926 [-5.3301 to 8.5152]
  Dyspnoea | 3.7134 [-0.3957 to 7.8226] | 0.5046 [-5.2542 to 6.2635]
  Insomnia | -2.6266 [-7.8402 to 2.5870] | -7.5026 [-14.8641 to -0.1411]
  Appetite loss | 13.7423 [9.9118 to 17.5727] | 10.9601 [5.6151 to 16.3051]
  Constipation | 8.0230 [3.9214 to 12.1246] | 4.0855 [-1.6913 to 9.8624]
  Diarrhoea | 6.0230 [2.9313 to 9.1147] | -0.1455 [-4.3834 to 4.0925]
  Financial Problems | 4.8435 [0.03603 to 9.6510] | 2.1140 [-4.7005 to 8.9284]
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Physical Functioning. Analysis of variance (ANOVA) included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.4975, ANOVA; Least Square (LS) Mean Difference = 2.1002, 95% CI 2-sided [-3.9855 to 8.1860]
Statistical Analysis 2: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Role Functioning. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.7600, ANOVA; LS Mean Difference = -1.4704, 95% CI 2-sided [-10.9358 to 7.9951]
Statistical Analysis 3: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Emotional Functioning. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.9949, ANOVA; LS Mean Difference = -0.02278, 95% CI 2-sided [-7.0350 to 6.9895]
Statistical Analysis 4: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Cognitive Functioning. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.6253, ANOVA; LS Mean Difference = -1.8213, 95% CI 2-sided [-9.1550 to 5.5125]
Statistical Analysis 5: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Social Functioning. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.7219, ANOVA; LS Mean Difference = 1.6126, 95% CI 2-sided [-7.2953 to 10.5205]
Statistical Analysis 6: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Global Health Status /QoL. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.2443, ANOVA; LS Mean Difference = 3.4989, 95% CI 2-sided [-2.4046 to 9.4023]
Statistical Analysis 7: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Fatigue. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.3287, ANOVA; LS Mean Difference = -3.3449, 95% CI 2-sided [-10.0739 to 3.3841]
Statistical Analysis 8: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Nausea/Vomiting. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.0485, ANOVA; LS Mean Difference = -4.1960, 95% CI 2-sided [-8.3635 to -0.02850]
Statistical Analysis 9: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Pain. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.0354, ANOVA; LS Mean Difference = -9.0950, 95% CI 2-sided [-17.5629 to -0.6271]
Statistical Analysis 10: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Dyspnoea. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.3724, ANOVA; LS Mean Difference = -3.2088, 95% CI 2-sided [-10.2784 to 3.8608]
Statistical Analysis 11: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Insomnia. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.2884, ANOVA; LS Mean Difference = -4.8760, 95% CI 2-sided [-13.9002 to 4.1482]
Statistical Analysis 12: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Appetite loss. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.4081, ANOVA; LS Mean Difference = -2.782, 95% CI 2-sided [-9.3926 to 3.8282]
Statistical Analysis 13: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Constipation. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.2750, ANOVA; LS Mean Difference = -3.9375, 95% CI 2-sided [-11.0245 to 3.1495]
Statistical Analysis 14: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Diarrhoea. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.0213, ANOVA; LS Mean Difference = -6.1685, 95% CI 2-sided [-11.4129 to -0.9241]
Statistical Analysis 15: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Financial Problems. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.5201, ANOVA; LS Mean Difference = -2.7295, 95% CI 2-sided [-11.0727 to 5.6137]

8. Secondary Outcome: Change From Baseline for EORTC QLQ Brain Neoplasm 20 (BN20) at Baseline, Post-Baseline (up to Month 30)
Description: EORTC QLQ-BN20 consisted of 20 items assessing visual disorders, motor dysfunction, communication deficit, various disease symptoms (e.g. headaches and seizures), treatment toxicities (e.g. hair loss) and future uncertainty. All of the 20 items are rated on a 4 point Likert scale from 1=not at all, 2=a little, 3=quite a bit and 4=very much, and were linearly transformed to a 0-100 scale, with higher scores indicating more severe symptoms.
Time Frame: Baseline, Post-Baseline (up to Month 30)
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
units on a scale
  Future uncertainty | -5.2779 [-9.2589 to -1.2968] | -8.5478 [-14.3337 to -2.7619]
  Visual disorder | -2.0869 [-4.5092 to 0.3354] | -3.202 [-6.7584 to 0.3528]
  Motor dysfunction | 5.4416 [2.3943 to 8.4888] | 6.5429 [2.1426 to 10.9433]
  Communication deficit | 4.7440 [1.6899 to 7.7980] | 4.6431 [0.2253 to 9.0609]
  Headaches | 4.3905 [0.6465 to 8.1345] | -3.9389 [-9.2879 to 1.4101]
  Drowsines | 11.7204 [7.6425 to 15.7983] | 8.2805 [2.3973 to 14.1637]
  Hair loss | 11.9235 [7.6344 to 16.2127] | 7.3328 [1.0111 to 13.6545]
  Itchy skin | 5.4882 [2.0875 to 8.8890] | 6.4690 [1.5048 to 11.4331]
  Weakness of legs | 8.9586 [4.9123 to 13.0048] | 7.9245 [2.0687 to 13.7804]
  Bladder control | 1.5020 [-1.0917 to 4.0957] | 1.9710 [-1.8122 to 5.7543]
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Future uncertainty. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.3613, ANOVA; LS Mean Difference = -3.2699, 95% CI 2-sided [-10.2983 to 3.7585]
Statistical Analysis 2: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Visual disorder. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.6146, ANOVA; LS Mean Difference = -1.1159, 95% CI 2-sided [-5.4654 to 3.2336]
Statistical Analysis 3: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Motor dysfunction. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.6860, ANOVA; LS Mean Difference = 1.1014, 95% CI 2-sided [-4.2449 to 6.4477]
Statistical Analysis 4: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Communication deficit. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.9706, ANOVA; LS Mean Difference = -0.1009, 95% CI 2-sided [-5.4680 to 5.2663]
Statistical Analysis 5: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Headaches. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.0124, ANOVA; LS Mean Difference = -8.3294, 95% CI 2-sided [-14.8550 to -1.8037]
Statistical Analysis 6: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Seizures. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.5997, ANOVA; LS Mean Difference = -1.0054, 95% CI 2-sided [-4.7654 to 2.7545]
Statistical Analysis 7: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Drowsiness. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.3458, ANOVA; LS Mean Difference = -3.4399, 95% CI 2-sided [-10.6002 to 3.7204]
Statistical Analysis 8: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Hair loss. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.2383, ANOVA; LS Mean Difference = -4.5908, 95% CI 2-sided [-12.2279 to 3.0464]
Statistical Analysis 9: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Itchy skin. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.7491, ANOVA; LS Mean Difference = 0.9807, 95% CI 2-sided [-5.0373 to 6.9988]
Statistical Analysis 10: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Weakness of legs. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.7755, ANOVA; LS Mean Difference = -1.0341, 95% CI 2-sided [-8.1508 to 6.0827]
Statistical Analysis 11: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Bladder control. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.8410, ANOVA; LS Mean Difference = 0.4690, 95% CI 2-sided [-4.1211 to 5.0591]

9. Secondary Outcome: Change From Baseline for Mini-Mental Status Examination (MMSE) at Baseline, Post-Baseline (up to Month 30)
Description: The MMSE briefly measures orientation to time and place, immediate recall, short-term verbal memory, calculation, language and construct ability. Each area tested had a designated point value, the total score can range from 0 to 30, with a higher score indicating better function.
Time Frame: Baseline, Post-Baseline (up to Month 30)
Population: ITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
units on a scale
  Orientation to time and place | -0.01771 [-0.1406 to 0.1052] | -0.2110 [-0.3907 to -0.03135]
  Immediate recall | -0.00264 [-0.02163 to 0.01635] | -0.03219 [-0.05888 to -0.00551]
  Repetitions required | -0.05763 [-0.1971 to 0.08180] | 0.08530 [-0.1212 to 0.2918]
  Calculations | -0.2153 [-0.3911 to -0.03952] | -0.2120 [-0.4706 to 0.04652]
  Short-term verbal memory | 0.2012 [0.1060 to 0.2964] | 0.1634 [0.02332 to 0.3034]
  Language and construct ability | -0.1254 [-0.2416 to -0.00908] | -0.2057 [-0.3765 to -0.03499]
  Total Score | -0.2871 [-0.7647 to 0.1905] | -0.5999 [-1.3069 to 0.1071]
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Orientation to time and place. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.0817, ANOVA; LS Mean Difference = -0.1933, 95% CI 2-sided [-0.4110 to 0.02438]
Statistical Analysis 2: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Immediate recall. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.0773, ANOVA; LS Mean Difference = -0.02955, 95% CI 2-sided [-0.06234 to 0.003241]
Statistical Analysis 3: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Repetitions required. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.2608, ANOVA; LS Mean Difference = 0.1429, 95% CI 2-sided [-0.1065 to 0.3924]
Statistical Analysis 4: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Calculations. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.9836, ANOVA; LS Mean Difference = 0.003262, 95% CI 2-sided [-0.3092 to 0.3158]
Statistical Analysis 5: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Short-term verbal memory. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.6610, ANOVA; LS Mean Difference = -0.03782, 95% CI 2-sided [-0.2071 to 0.1315]
Statistical Analysis 6: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Language and construct ability. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.4464, ANOVA; LS Mean Difference = -0.08037, 95% CI 2-sided [-0.2875 to 0.1268]
Statistical Analysis 7: Comparison: Bevacizumab + Irinotecan vs Temozolomide; Total score. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.4717, ANOVA; LS Mean Difference = -0.3128, 95% CI 2-sided [-1.1658 to 0.5402]

10. Secondary Outcome: Change From Baseline for Karnofsky Performance Status (KPS) Score at Baseline, Post-Baseline (up to Month 30)
Description: KPS is an 11-level score (0, 10, 20, 30, 40, 50, 60, 70, 80, 90, and 100) which ranges between 0 (death) to 100 (complete healthy status); a higher score represents a higher ability to perform daily tasks. Deterioration in KPS was defined as decrease of 20 or more points in KPS score.
Time Frame: Baseline, Post-Baseline (up to Month 30)
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 54
units on a scale | -3.3399 [-5.2132 to -1.4666] | -5.4909 [-8.2693 to -2.7126]
Statistical Analysis 1: Comparison: Bevacizumab + Irinotecan vs Temozolomide; KPS score. ANOVA included all post-baseline data (Months 3 through 21); Test type: Superiority or Other; p = 0.2078, ANOVA; LS Mean Difference = -2.1510, 95% CI 2-sided [-5.4983 to 1.1963]

11. Secondary Outcome: Percentage of Participants Who Received Corticosteroid for Glioblastoma
Description: Participants used corticosteroids for the glioblastoma condition. Corticosteroids included dexamethasone, methylprednisone, fortecortin, hydrocortisone, urbason, and prednisolone.
Time Frame: From baseline to Month 6
Population: The safety population (SAF) was defined to include all participants who received at least 1 dose of study medication. Data were analyzed according to the treatment actually received (as treated).
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 119 | 55
percentage of participants | 80.0 | 78.7

12. Secondary Outcome: Time to Treatment Failure
Time Frame: From baseline until end of study (up to 4.5 years)
Population: Data for this outcome measure were not collected as this outcome was removed as per changes in planned analysis.
Measure: Median (Full Range); unit: years
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Number analyzed (Participants) | 116 | 55
years | NA [NA to NA] — Data for time to treatment failure were not collected as this outcome was removed as per changes in planned analysis | NA [NA to NA] — Data for time to treatment failure were not collected as this outcome was removed as per changes in planned analysis

ADVERSE EVENTS:
Time Frame: 4 years, 5 months,24 days
Groups:
- Temozolomide: In the Concurrent Phase participants received radiotherapy in daily fractions of 1.8 to 2 Gy given 5 fractions per week for 6 to 7 week and temozolomide (TMZ) capsule 75 mg/m^2 BSA daily from the first day to the last day of radiotherapy . There was a 4 week treatment break. Participants then entered the Maintenance Phase where they received six 28-day cycle of TMZ 150 to 200 mg/m^2 BSA daily in the first 5 days of each cycle until PD or for a maximum treatment period of 2 years after inclusion of the last participant. Only participants with progressive disease during or after TMZ therapy could receive bevacizumab (BEV)/irinotecan (IRI) or BEV monotherapy as optional second-line study therapy at the discretion of the investigator or and, if eligible.
Arm/Group | Bevacizumab + Irinotecan | Temozolomide
Serious Adverse Events (participants affected / at risk) | 86/119 | 46/55
Other Adverse Events (participants affected / at risk) | 107/119 | 37/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Irinotecan (N=119) | Temozolomide (N=55)
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 5
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Diverticular perforation (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 41 | 20
Hernia (General disorders) | 1 | 0
Impaired healing (General disorders) | 2 | 2
Local swelling (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 2
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
extradural abscess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 3 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 3 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 3
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 4
Cerebral cys (Nervous system disorders) | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Coma (Nervous system disorders) | 0 | 1
Complex partial seizures (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 17 | 9
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 6 | 6
Grand mal convulsion (Nervous system disorders) | 5 | 1
Headache (Nervous system disorders) | 2 | 4
Hemiparesis (Nervous system disorders) | 1 | 4
Hemiplegia (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Intracranial haematoma (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 2 | 3
Postictal paralysis (Nervous system disorders) | 2 | 0
Status epilepticus (Nervous system disorders) | 2 | 0
Subdural hygroma (Nervous system disorders) | 1 | 2
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Cystitis glandularis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Therapeutic procedure (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Irinotecan (N=119) | Temozolomide (N=55)
Diarrhoea (Gastrointestinal disorders) | 54 | 8
Nausea (Gastrointestinal disorders) | 88 | 28
Headache (Nervous system disorders) | 60 | 22

LIMITATIONS AND CAVEATS:
Data for time to treatment failure were not collected as this outcome was removed as per changes in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.